CLINICAL TRIAL: NCT01411566
Title: Evaluation of an Integrative Therapeutic Concept for Schizophrenic Patients With Comorbid Substance Use Disorder
Brief Title: Clinical Intervention Psychosis and Addiction
Acronym: KLIPS
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Dr. Joerg Daumann, PhD, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Koeln-Fortune 104/2010
Record Dates: First submitted 2011-03-02; First posted 2011-08-08 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-02

CONDITIONS: Psychosis; Substance Abuse
Keywords: KLIPS
MeSH Terms: conditions — Psychotic Disorders; Substance-Related Disorders | interventions — mica

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Behavioral: Skills trainig for patients with dual diagnosis
- Control (Active Comparator)
  Interventions: Behavioral: regular treatment

INTERVENTIONS:
Behavioral: Skills trainig for patients with dual diagnosis — Skills trainig for patients with dual diagnosis
  Arms: Treatment
Behavioral: regular treatment — regular treatment
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate an integrative therapeutic concept for schizophrenic patients with comorbid substance use disorder.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia
* Addiction
* Written statement of agreement
* Majority

Exclusion Criteria:

* Acute psychosis
* Further neuropsychiatric disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-11 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Substance use | one year
Substance use | 3 months
Substance use | 6 months
Change in drug use motivation | 3 months
Change in drug use motivation | 6 months
Change in drug use motivation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Daumann, PhD, Study Chair — University of Cologne
Locations (1):
- LVR Clinic Cologne - Academic Clinic of the University of Cologne, Cologne, Germany